CLINICAL TRIAL: NCT06322537
Title: Albumin Utilization for Intravascular Volume Replacement in Adult Cardiac Surgical Patients : A Multi-centre, Retrospective, Cohort Study
Brief Title: Albumin Utilization in Adult Cardiac Surgical Patients: Retrospective
Acronym: AlbACS-1R
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kingston Health Sciences Centre (Other); Unity Health Toronto (Other); McMaster University (Other); Sunnybrook Health Sciences Centre (Other); London Health Sciences Centre (Other); The Ottawa Hospital (Other); Vancouver General Hospital (Other); Royal Columbian Hospital Foundation (Other); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5339
Record Dates: First submitted 2024-02-21; First posted 2024-03-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Surgical Procedures; Albumin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Adult (≥18 years old) patients who have undergone cardiac surgery.

SUMMARY:
All heart surgery patients universally require hydration, which is given through a vein in the arm, but practices for treating patients are not universal. There are disagreements about whether crystalloids should be used alone or in combination with albumin. This question has important implications because albumin is an expensive blood product in relatively limited supply, and 20% of its use is by heart surgery patients. The goal of this study is to learn more about how crystalloids and albumin are used during heart surgery, as well as, key patient outcomes.

DETAILED DESCRIPTION:
The goal of this proposed multicentre retrospective cohort study is to characterize perioperative usage patterns of crystalloids and albumin, as well as key patient outcomes, in cardiac surgical patients. This study will also address numerous other knowledge gaps in the area of perioperative blood product management and fluid administration in cardiac surgery and define a collaborative group to support future research in this field.

The primary objective is to obtain granular information on if, when, and how albumin is given perioperatively to cardiac surgical patients. This includes the doses and settings in which albumin is used, the types of crystalloid solutions (balanced or unbalanced) used, and when albumin is used (for example, while on cardio-pulmonary bypass, in the ICU, or on the ward) in perioperative cardiac surgical care across institutions. This important information about the scope of albumin and crystalloid use across the country will inform the design of our future intervention and control arms in the planned definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Cardiac surgery with the use of cardiopulmonary bypass
* Cardiac surgery without the use of cardiopulmonary bypass

Exclusion Criteria

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include up to 500 adult (≥18 years old) patients who have undergone major cardiac surgery. All adult (≥18 years old) patients who have undergone cardiac surgery (with or without the use of cardio-pulmonary bypass) will be eligible. There are no specific exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 505 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Albumin | On CPB, in the operating room but not during CPB, in the ICU, on the ward to post operative day 28.
  Type, dose and timing of administration, the setting in which it was ordered, indication for use, and the type of provider responsible for the patient at administration (surgeon, anesthesiologist, intensivist, nurse practitioner).
Crystalloid, volume dose and type administered | On CPB, in the operating room but not during CPB, in the ICU, on the ward to post operative day 28.
  Type and volume of crystalloid given (Normal saline, Ringer's Lactate, Plasmalyte-148, and others), as well as the setting of administration will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD MSc FRCPC, Principal Investigator — Toronto General Hospital - University Health Network
Locations (10):
- Canada (10):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Science Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No